CLINICAL TRIAL: NCT07016269
Title: Multi-center, Randomized, Double-blind, Placebo Controlled, Parallel Clinical Trial for the Evauation of the Efficacy and Safety of CnU Cap. 500 mg in Patients With Biliary Dyspepsia
Brief Title: A Study to Evaluate the Efficacy and Safety of CnU Cap. 500 mg in Patients With Biliary Dyspepsia
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Myungmoon Pharma. Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MMP-402
Record Dates: First submitted 2025-05-29; First posted 2025-06-11 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Biliary Dyspepsia
MeSH Terms: interventions — 1-(2-chloroethyl)-1-nitrosourea

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CnU capsule 500 mg(250mg 2 capsule) (Experimental)
  Interventions: Drug: CnU capsule 500 mg(250mg 2 capsule)
- CnU placebo capsule 500 mg(250mg 2 capsule) (Placebo Comparator)
  Interventions: Drug: CnU placebo capsule 500 mg(250mg 2 capsule)

INTERVENTIONS:
Drug: CnU capsule 500 mg(250mg 2 capsule) — According to the randomly assigned treatment groups, the medication will be administered orally at a dose of 500 mg (2 capsules) once daily for a total of 24 weeks, preferably at the same time each day after meals.
  Arms: CnU capsule 500 mg(250mg 2 capsule)
Drug: CnU placebo capsule 500 mg(250mg 2 capsule) — According to the randomly assigned treatment groups, the medication will be administered orally at a dose of 500 mg (2 capsules) once daily for a total of 24 weeks, preferably at the same time each day after meals.
  Arms: CnU placebo capsule 500 mg(250mg 2 capsule)

SUMMARY:
The objective of this clinical trial is to evaluate the efficacy and safety of CnU capsule 500 mg administration in patients with biliary dyspepsia

ELIGIBILITY:
[Inclusion Criteria]

1. Individuals who have voluntarily agreed to participate in this clinical trial
2. Adults aged 19 years and older
3. Individuals with pain localized to the epigastrium and/or right upper quadrant, as defined by the ROME IV diagnostic criteria

   * Rome IV criteria(Functional gallbladder and sphincter of Oddi disorders Diagnostic criteria) 1) Builds up to a steady level and lasts 30 minutes or longer 2) Occurring at different intervals (not daily) 3) Severe enough to interrupt daily activities or lead to an emergency department visit 4) Not significantly (<20%) related to bowel movements 5) Not significantly (<20%) relieved by postural change or acid suppression
   * Supportive criteria:

The pain may be associated with:

1) Nausea and vomiting 2) Radiation to the back and/or right infrasubscapular region 3) Waking from sleep

4. Individuals without any organic lesions on abdominal ultrasonography performed during screening that could explain biliary colic symptoms due to gallstones

[Exclusion Criteria]

1. Medical History

1. Patients with frequent biliary colic or biliary tract infections (e.g., severe pancreatic changes such as ileal resection, surgery, or partial ileitis, which may alter the composition of enterohepatic bile acid circulation).
2. Patients with obstructive jaundice.
3. Patients with liver disease.
4. Patients with severe renal disease.
5. Patients with severe biliary obstruction (due to the potential choleretic effect, symptoms may worsen).
6. Patients with underlying conditions that may worsen biliary obstruction (e.g., cholangiocarcinoma, cholangitis, biliary cysts).
7. Patients with acute cholecystitis.
8. Patients with a clear etiology of dyspepsia (e.g., those with endoscopically or clinically confirmed GI abnormalities such as gastric ulcer, gastroparesis; regular NSAID users; or those with prominent heartburn).
9. Patients with peptic ulcer disease (due to the potential for mucosal irritation and symptom aggravation).
10. Patients with inflammatory bowel diseases such as Crohn's disease.
11. Patients with cholestasis.
12. Patients with abnormal gallbladder contractility.
13. Patients with a history of malignancy within 5 years prior to screening.
14. Patients with a history of gastrointestinal surgery.
15. Patients known to be hypersensitive to any components or excipients of the investigational product.
16. Patients with clinically significant disorders of the cardiovascular, gastrointestinal, respiratory, endocrine, or central nervous systems, or with a history or presence of psychiatric illness that may significantly affect participation in the study.
17. Individuals with a history of drug or alcohol abuse.

2. Abnormal Laboratory Findings at Screening

1. Body Mass Index (BMI) ≥ 35 kg/m².
2. ALT or AST > 2.0 × upper normal limit (UNL).
3. Total bilirubin > 2.0 × UNL.
4. Estimated glomerular filtration rate (eGFR) < 60 mL/min/1.73 m² (based on the CKD-EPI equation).
5. Positive serologic test results for any of the following:

   - Hepatitis B surface antigen (HBsAg)
   * Hepatitis C antibody (HCV Ab)
   * Human immunodeficiency virus antibody (HIV Ab)
   * Syphilis reagin test

     3. Prohibited Concomitant Medications and Therapies

Subjects taking the following medications must undergo the specified washout period before enrollment:

1. Within 1 week prior to screening: Drugs that stimulate bile secretion (e.g., estrogens, hormonal contraceptives, certain lipid-lowering agents) Drugs that reduce blood cholesterol (e.g., clofibrate)
2. Within 2 weeks prior to screening: Cholestyramine, colestipol, activated charcoal, or antacids containing magnesium or aluminum hydroxide
3. Within 4 weeks prior to screening: Oral gallstone-dissolving agents such as chenodeoxycholic acid (CDCA), ursodeoxycholic acid (UDCA), HMG-CoA reductase inhibitors, or terpene-based drugs
4. Within 4 weeks prior to screening: Bile acid therapies

   The following medication is strictly prohibited, regardless of washout period:
   * Alpha-methyldopa

     4. Pregnant or lactating women will be excluded from the study.

     5. Contraception

   Subjects or their partners who are not using medically acceptable methods of contraception throughout the study period will be excluded. Acceptable methods include:

1) Proven intrauterine devices (IUD) or intrauterine systems (IUS) 2) Dual barrier methods (e.g., male condom with diaphragm or cervical cap, used with a spermicide) 3) Permanent sterilization (e.g., vasectomy, tubal ligation, salpingectomy, or hysterectomy)

6. Other Individuals deemed by the investigator to be unsuitable for participation in this clinical trial for any reason.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 358 (Estimated)
Dates: Start 2025-08-29 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Symptom improvement rate at Week 24 using the Global Overall Symptom Scale (GOS) in patients with biliary dyspepsia | Baseline and Week 24
  * Description: The Global Overall Symptom Scale assesses the overall severity of upper abdominal symptoms such as pain or discomfort, bloating, excessive belching, and nausea. Symptoms are rated on a 7-point Likert scale, where 1 = no symptoms and 7 = very severe symptoms.
  * Outcome Definition: Improvement is defined as a decrease of 2 or more points compared to baseline.
  * Unit of Measure: Percentage of participants with ≥2-point reduction

SECONDARY OUTCOMES:
1. Symptom improvement rate using the GOS in patients with biliary dyspepsia 2. Change in dyspepsia symptom scores using the NDI-K 3. Change in quality of life scores using the NDI-K | Baseline, Week 4, Week 12, and Week 24
  1. Symptom improvement rate at Weeks 4 and 12 using the GOS in patients with biliary dyspepsia
     * Time Frame: Baseline, Week 4, and Week 12
     * Description: The GOS evaluates upper abdominal symptoms using a 7-point Likert scale, where 1 = no symptoms and 7 = very severe symptoms.
     * Outcome Definition: Improvement is defined as a decrease of 2 or more points compared to baseline.
     * Unit of Measure: Percentage of participants with ≥2-point reduction
  2. Change in dyspepsia symptom scores from baseline using the NDI-K
     * Time Frame: Baseline, Week 4, Week 12, and Week 24
     * Outcome Definition: Change in total and subscale scores from baseline.
     * Unit of Measure: Mean change in score
  3. Change in quality of life scores from baseline using the NDI-K QoL subscale
     * Time Frame: Baseline, Week 4, Week 12, and Week 24
     * Outcome Definition: Change in QoL subscale scores from baseline
     * Unit of Measure: Mean change in score

CONTACTS AND LOCATIONS:
Locations (6):
- South Korea (6):
  - Pusan National University Hospital, Busan
  - CHA Bundang Medical Center, Gyeonggi-do
  - Hallym University Dongtan Sacred Heart Hospital, Gyeonggi-do
  - Soonchunhyang University Cheonan Hospital, Gyeonggi-do
  - Inha University Hospital, Incheon
  - Gangnam Severance Hospital, Seoul